CLINICAL TRIAL: NCT04178707
Title: Intervention With Microdialysis Measurements in Anal Fistula
Brief Title: Anal Fistula and Microdialysis - What is Yet to Learn?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Umeå (Other)
Responsible Party: Principal Investigator, Karin Gustafsson, Medical Doctor, Principal Investigator, University Hospital, Umeå
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UMUmea
Record Dates: First submitted 2019-10-25; First posted 2019-11-26 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: Microdialysis is used to investigate the inner enviorment of anal fistulas. The patient will be its own control with measurements at prior to intervention and after operative procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Using microdialysis the patients inner enviorment of the anal fistula will be measured - levels of lactate, glucose and pyruvate.
  Interventions: Device: OnZurf Probe, Senzime AB, Uppsala, Sweden

INTERVENTIONS:
Device: OnZurf Probe, Senzime AB, Uppsala, Sweden — Probe is inserted into the fistula and measurements are made of the inner environment.

SUMMARY:
Anal Fistula can be a challenging condition to treat. Microdialysis has never before been used to examine the inner environment of anal fistula. This is now going to be performed.

DETAILED DESCRIPTION:
Patients with anal fistula can have a reduced quality of life for years do to fistula complications. This condition is not well researched and more knowledge is needed to provide better care. Microdialysis has been used to study other organs of the body such as the brain, liver and GI-tract. Upcoming study is going to study the inner environment of the anal fistula in regards to lactate, pyruvate and glucose.

The study group is patients with anal fistula that with a need for seton treatment. Measurements with microdialysis will take place before operative procedure and one month after getting their seton inserted.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* to be able to understand and accept the terms of study

Exclusion Criteria:

* age under 18
* dementia, language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
measurements of glucose in anal fistula using microdialysis | baseline measurement, 1 month follow up
  measurements of glucose in fistula using microdialysis, change in value is being assessed

SECONDARY OUTCOMES:
measurement of pyruvate in anal fistula using microdialysis | baseline measurement, 1 month follow up
  measurement of pyruvate measurements in fistula using microdialysis, change in value is being assessed

OTHER OUTCOMES:
measurement of lactate in anal fistula using microdialysis | baseline measurement, 1 month follow up
  measurement of lactate in fistula using microdialysis, change in value is being assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Gunnarsson, Professor, Study Chair — University Hospital, Umeå
Locations (1):
- Umea University Hospital, Umeå, Västerbotten County, Sweden